CLINICAL TRIAL: NCT00755820
Title: Food Exposure Therapy in Anorexia Nervosa
Status: Completed | Type: Observational
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: The Hilda & Preston Davis Foundation (Other); National Alliance for Research on Schizophrenia and Depression (Other)
Responsible Party: Sponsor
Other Study IDs: 5457
Record Dates: First submitted 2008-09-18; First posted 2008-09-19 (Estimated); Last update posted 2012-10-26 (Estimated); Status verified 2012-10

CONDITIONS: Anorexia Nervosa
MeSH Terms: conditions — Anorexia Nervosa | interventions — Implosive Therapy; Cycloserine

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- EXP-DCS/Exposure-D-cycloserine: Exposure Therapy + D-Cycloserine
  Interventions: Behavioral: Exposure Therapy + D-Cycloserine
- EXP-PBO: Exposure Therapy + Placebo
  Interventions: Behavioral: Exposure Therapy + Placebo
- SP: Supportive psychotherapy
  Interventions: Behavioral: Supportive Psychotherapy

INTERVENTIONS:
Behavioral: Exposure Therapy + D-Cycloserine — Exposure therapy with d-cycloserine medication
  Groups: EXP-DCS/Exposure-D-cycloserine
Behavioral: Exposure Therapy + Placebo — Exposure therapy with placebo medication
  Groups: EXP-PBO
Behavioral: Supportive Psychotherapy — Supportive psychotherapy
  Groups: SP

SUMMARY:
This is a research study to determine whether a medication called D-cycloserine (DCS) in combination with a type of psychotherapy called Exposure Therapy is helpful to patients with anorexia nervosa.

DETAILED DESCRIPTION:
This is a research study to determine whether a medication called D-cycloserine (DCS) in combination with a type of psychotherapy called Exposure Therapy is helpful to patients with anorexia nervosa. DCS is approved by the FDA as an antibiotic medication, but has not been approved by the FDA for the treatment of anorexia nervosa. Past studies have found that DCS together with Exposure Therapy can help people with height phobia, social phobia, and obsessive compulsive disorder. Anorexia nervosa often includes phobia-like fears, obsessive thoughts, and compulsive rituals, so the current study aims to determine whether DCS paired with Exposure Therapy can also help people with anorexia nervosa. Anorexia nervosa is a disorder characterized by self-starvation, extreme weight loss, and difficulty maintaining a normal weight. You have been asked to participate in this study because you have been given a diagnosis of anorexia nervosa. In this study you will receive one of three therapies: Exposure Therapy with DCS, Exposure Therapy with placebo (inactive medication), or Treatment as Usual. You will participate in a total of four test meals in a laboratory setting. A total of 70 individuals with anorexia nervosa will participate in this study. Twenty individuals who have never had an eating disorder will participate in one portion of this study.

ELIGIBILITY:
Inclusion Criteria for Patients:

* DSM-IV-TR™ diagnosis of anorexia nervosa (restricting or binge-purge subtype) on admission
* Subjects will have achieved 90% of ideal body weight (IBW)
* Age 18-45
* Medically stable
* Participation in inpatient treatment
* Subjects must have signed informed consent document indicating that they understand the purpose of and procedures required for the study and are willing to participate in the study.

Exclusion Criteria for Patients:

* Any other current major Axis I disorder, except OCD or MDD (mild)
* On psychotropic medication, including benzodiazepines (At the start of the study, subjects will be free of fluoxetine for 4 weeks, and free of all other medications for a minimum of 2 weeks.)
* History of a seizure disorder
* Abnormal liver function
* Renal insufficiency
* Known hypersensitivity to D-cycloserine
* Pregnant or lactating
* Acute suicidality (suicidality or self injury in the last 3 months)

Inclusion Criteria for Healthy Controls:

* BMI ≥ 19.0 kg/m2
* Age 18-45 years
* Subjects must have signed informed consent document indicating that they understand the purpose of and procedures required for the study and are willing to participate in the study.

Exclusion Criteria for Healthy Controls:

* Current Major Axis I disorder (including Eating Disorder, Major Depression,Bipolar Disorder, Schizophrenia, Substance Abuse/Dependence) History of an Eating Disorder
* Current use of psychotropic medication or other medication known to affect mood and/or anxiety (e.g. b-agonist inhalers, oral steroids)
* Major medical condition

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Inpatients receiving treatment for anorexia nervosa
Sampling Method: Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2008-01; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joanna Steinglass, M.D., Principal Investigator — CUMC/NYSPI
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

REFERENCES:
- [Derived] Steinglass JE, Sysko R, Mayer L, Berner LA, Schebendach J, Wang Y, Chen H, Albano AM, Simpson HB, Walsh BT. Pre-meal anxiety and food intake in anorexia nervosa. Appetite. 2010 Oct;55(2):214-8. doi: 10.1016/j.appet.2010.05.090. Epub 2010 Jun 4. PMID 20570701